CLINICAL TRIAL: NCT02978937
Title: Obstrutive Sleep Apnea: is it a Biomarker of Metabolically Healthy vs. Unhealthy Obese
Brief Title: Obstructive Sleep Apnea and Metabolic Health
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, David Bradley MD, MD, Ohio State University
Other Study IDs: 2015E0155
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Sleep; Apnea; Metabolism Disorder
MeSH Terms: conditions — Sleep Apnea Syndromes; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metabolically healthy and abnormal obese: Obese patients divided into two groups according to their metabolic profile (healthy vs unhealthy)

SUMMARY:
This is an observational study involving chart review of patients seen in the bariatric clinic since 2012 at The Ohio State University (OSU). Obese patients will be divided into two groups according to their metabolic profile (healthy vs unhealthy). The assignment to each group will be determined by the presence of diagnosis of hypertension, diabetes mellitus and/or dyslipidemia. The presence of at least 2 diagnoses will be defined as metabolically unhealthy. Then, each group will be divided based on the presence of Obstructive Sleep Apnea diagnosis. All data will be collected through a review of the patient's electronic medical record from the bariatric clinic database (the investigators will collect variables as age, gender, race, BMI, smoking status, the presence of diagnosis as Obstructive sleep apnea, hypertension, diabetes, hyperlipidemia). The investigators will analyze that data and establish if there is any correlation between sleep apnea and the subjects' metabolic profile.

DETAILED DESCRIPTION:
Obesity is associated with numerous metabolic complications including Type 2 diabetes mellitus, hypertension, dyslipidemia, cardiovascular disease (CVD) and several forms of cancer. However, the presence of these obesity-related metabolic abnormalities varies among obese individuals. The phenotype of a metabolically healthy obese (MHO) individual was initially described in 1980 and includes a subset of obese patients (as defined by BMI) who do not manifest the typical metabolic abnormalities associated with obesity. Although results are conflicting and highly dependent on patient population and diagnostic criteria for metabolic health, these individuals tend to have a preserved level of insulin sensitivity, absence of hypertension, and a more favorable lipid, inflammatory, hormonal, hepatic, and immunologic profile compared to the majority of metabolically abnormal obese (MAO) patients. This seeming paradox underscores that excess body the weight is not the sole determinant of obesity-related complications and allows for novel pathogenic investigation.

The postulated mechanism(s) underlying the differential metabolic profile in these individuals is not well known and the physiologic and molecular basis for 'healthy' obesity remains relatively undiscovered. In addition, a recent meta-analysis demonstrated that although MHO patients have a comparable metabolic profile to normal the weight individuals, their risk of adverse, long-term CV and mortality outcomes remains higher, calling into question the clinical importance of the healthy obese categorization. Despite these knowledge gaps, a limited number of studies have recently attempted to elucidate the processes that lead to the MHO profile, including characterization of lifestyle factors, adipocyte size, amount and location of ectopic fat, inflammatory mediators, and immune cells, and differences in gene expression.

The prevalence of obstructive sleep apnea (OSA) increases with increasing BMI and has also been linked to various cardiometabolic abnormalities. Patients with OSA experience repetitive episodes of hypoxia and reoxygenation during transient cessation of breathing that may provoke adverse systemic effects. These effects are reflected in increased levels of biomarkers linked to endocrine-metabolic and cardiovascular disease. OSA may exert negative effects on the cardiovascular system through multiple mechanisms including hypoxemia, sleep disruption, activation of the sympathetic nervous system, and inflammatory activation. In spite of this connection, the contribution of these deleterious effects in determining the phenotype of an obese patient (MHO vs. MAO) is unknown. Furthermore, the prevalence of OSA in these two subsets is not the well established.

In this study, the investigators hypothesize the prevalence of OSA is higher in MAO compared to BMI-matched MAO patients

Aim 1:

Define the prevalence of OSA in metabolically-healthy obese and metabolically abnormal obese (MHO and MAO) patients.

Aim 2:

Elucidate the association of OSA disease severity parameters with markers of clinically available abnormal metabolic profile (elevated cholesterol, blood pressure, fasting glucose/hemoglobin A1c, inflammatory markers, and insulin resistance if available).

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 88 year old
* BMI ≥ 30 kg/m2

Exclusion Criteria:

◦ Lack of pertinent clinical data to include in the study.

Ages: 21 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include a representative sample of the patient population at OSU, which is 59% Caucasian, 39% African American, and the remainder of mixed, Asian, or Native American descent. The investigators will review outpatient data from subjects seen at OSU Wexner Medical Center for Minimally Invasive surgery. The individual cohorts will then be divided based on the presence of OSA and metabolic abnormalities.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-11 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Define the prevalence of OSA in metabolically-healthy obese and metabolically abnormal obese (MHO and MAO) patients. | 2 years
Elucidate the association of OSA disease severity parameters with markers of clinically available abnormal metabolic profile | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Bradley, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Publications